CLINICAL TRIAL: NCT03896334
Title: Effect of Isometric Handgrip Training on Ambulatory Blood Pressure: a Multi-center Study
Brief Title: Effect of Isometric Handgrip Training on Ambulatory Blood Pressure in Patients With Hypertension
Acronym: ISOPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Aline Mendes Gerage, Principal Investigator, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISOPRESS_MULTICENTER STUDY
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric handgrip training (Experimental): All participants that will be assigned to supervised isometric handgrip training will train three times per week, during 24 weeks. They will perform a bout of isometric handgrip exercise: four sets of 2-min of isometric contractions (using alternate hands) at 30% of maximal voluntary contraction.
  Interventions: Behavioral: Supervised Isometric Handgrip Training
- Control group (Sham Comparator): All participants randomized to control group will realize stretching and relaxation exercises, three times per week, during 24 weeks.
  Interventions: Behavioral: Sham comparator - stretching and relaxation exercises

INTERVENTIONS:
Behavioral: Supervised Isometric Handgrip Training — The participants randomized to the experimental group will perform 24 weeks of isometric handgrip exercise training, three times/week for 16 minutes with time to rest.
  Arms: Isometric handgrip training
Behavioral: Sham comparator - stretching and relaxation exercises — The participants randomized to the control group (active comparator) will perform 24 weeks of stretching and relaxation exercise training, three times/week for 16 minutes with time to rest.
  Arms: Control group

SUMMARY:
Meta-analysis studies have demonstrated that isometric training with handgrip promotes reductions in clinical blood pressure, reaching 8 mmHg for systolic blood pressure and 4 mmHg for diastolic. However, the effects of this training modality on ambulatory blood pressure, which is better discriminant of cardiovascular risk than clinical BP, remains uncertain. Thus, the ISOPRESS Network, consists of researchers from Brazilian institutions of education and research (Federal University of Santa Catarina, Federal University of Amazonas, Federal University of Sergipe, Federal Rural University of Pernambuco and Universidade Nove de Julho), will conduct a multi-center study to analyze the effects of isometric handgrip training on clinic and 24-h ambulatory blood pressure in patients with hypertension. For this, each research center will conduct a randomized controlled trial with medicated patients with hypertension, of both sex. The participants will be randomized into two groups: isometric handgrip training group (HBT: n = 25 per center) and control group (CG: n = 25 per center).Subjects assigned to the HBT will train three times per week, four sets of 2-min isometric contractions (using alternate hands) at 30% of maximal voluntary contraction, during 24 weeks. Subjects randomized to the CG will perform stretching and relaxation exercises three times per week, during 24 weeks. The evaluations will occur in three moments: baseline, post-12 and post-24 weeks. The primary outcome will be ambulatory blood pressure, while clinic blood pressure and cardiac autonomic modulation will be analyzed as secondary outcomes. For data analysis, in addition to descriptive statistics, two-way ANOVA for mixed model will be applied for within and between groups comparison. The level of significance that will be adopted is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension, controlled by up to three antihypertensive medications
* Blood pressure levels between 130 and 180 mmHg
* No high cardiovascular risk (no other cardiovascular, metabolic or pulmonary disease nor any signals or symptoms of these disease)
* Not engaged in a physical exercise program for at least six months
* Not present cognitive impairment (Montreal Cognitive Assessment ≥ 26 points)

Exclusion Criteria:

* Adherence to less than 85% of training sessions
* Diagnosis of other cardiovascular diseases or diabetes during the course of the study
* Adherence to another supervised physical exercise program
* Change in medication class and/ or dose during the study
* Aggravation of the disease (i.e. blood pressure above 180 or use of four or more medications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in ambulatory systolic blood pressure | Baseline, 12 weeks 24 weeks
  24h-ambulatory blood pressure monitoring
Change in ambulatory diastolic blood pressure | Baseline, 12 weeks 24 weeks
  24h-ambulatory blood pressure monitoring
Change in ambulatory mean blood pressure | Baseline, 12 weeks 24 weeks
  24h-ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Change in clinic systolic blood pressure | Baseline, 12 weeks 24 weeks
  Clinic blood pressure will be checked using an automatic instrument
Change in clinic diastolic blood pressure | Baseline, 12 weeks 24 weeks
  Clinic blood pressure will be checked using an automatic instrument
Change in clinic mean blood pressure | Baseline, 12 weeks 24 weeks
  Clinic blood pressure will be checked using an automatic instrument
Change in heart rate variability | Baseline, 12 weeks 24 weeks
  For heart rate variability assessment, R-R interval will be obtained using a heart rate monitor (POLAR, RS 800CX), following the recommendations of the Task Force of the European Society of Cardiology and the North American.

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina
  - Federal University of Sergipe, Aracaju
  - Federal University of Amazonas, Parintins
  - Federal Rural University of Pernambuco, Recife
  - Universidade Nove de Julho, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided